CLINICAL TRIAL: NCT04420494
Title: Umbilical Cord Blood Treatment for Refractory Immune Cytopenia: a Single-arm Prospective Study
Brief Title: Umbilical Cord Blood Treatment for Refractory Immune Cytopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2433
Record Dates: First submitted 2020-04-27; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Umbilical Cord Blood; Refractory Immune Cytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with umbilical cord blood (Experimental)
  Interventions: Other: Umbilical Cord Blood

INTERVENTIONS:
Other: Umbilical Cord Blood — The diagnosis is definitely immune cytopenia (IRC), including autoimmune hemolytic anemia (AIHA, Hgb <100g / L, acquired pure red aplastic anemia (PRCA, Hgb <100g / L, EVANS syndrome , Hgb <100g / L and / or platelet count <30 × 109 / L, or blood cell reduction secondary to immune diseases (the same as the treatment indications, or neutrophils <0.5 × 109 / L), at least after hormone therapy Patients who are ineffective (did not reach PR after 4 weeks of hormone therapy) or who have not achieved PR after 3-5 mg / kg / d of cyclosporine. These patients would be treated with umbilical cord blood.

SUMMARY:
Immune-related hematocytopenia is a type of immunity Inflammatory cytopenia-mediated diseases, hormones and immunosuppressants are its first-line treatment. However, conventional immunosuppressants are ineffective or have a high recurrence rate. And some patients are not effective for these treatments, due to infection of blood cells, bleeding, decreased quality of life, and even severe death. There is currently no effective method for such patients. This study intends to recruit IRIC patients, give cord blood infusion, observe its efficacy and safety, and detect changes in inflammation-related indicators before and after treatment. There are no relevant reports at China and abroad. This study can provide new treatment options for patients with IRIC.

DETAILED DESCRIPTION:
Immune-related hematocytopenia (IRC- autoimmune hemolytic anemia (AIHA), Evans syndrome, acquired acquired pure red aplastic anemia (PRCA), autoimmune disease with cytopenia, etc.) is a type of immunity Inflammatory cytopenia-mediated diseases, hormones and immunosuppressants are its first-line treatment. However, conventional immunosuppressants are ineffective or have a high recurrence rate, known as refractory immune-related cytopenia (IRIC). Subsequent other second-line treatments such as other immunosuppressive agents, CD20 monoclonal antibodies, anti-human lymphocyte immunoglobulin (ATG ), And even splenectomy have problems such as high side effects, high price, slow onset of effect, and low efficiency. And some patients are not effective for these treatments, due to infection of blood cells, bleeding, decreased quality of life, and even severe death. There is currently no effective method for such patients.

Studies have shown that certain factors induce the loss of autoimmune tolerance in IRC patients, and the autoantigens of bone marrow hematopoietic cells are presented by dendritic cells, stimulating T cells, resulting in B cell activation and hyperfunction to produce specific autoantibodies; among them, helper T cells ( Th) Abnormal activation of 17 and follicular helper T cells (Tfh), the negative regulatory function of regulatory T cells and regulatory B cells weakens, and also promotes the production of autoantibodies. However, the bone marrow hematopoietic function caused by autoantibodies destroying or inhibiting hematopoietic cells is low or ineffective. Studies have pointed out that hematopoietic therapy is the key to curative treatment. At present, the safety and effectiveness of umbilical cord blood in the treatment of malignant / non-malignant hematological diseases have been confirmed and are widely used. In non-myeloablative therapy, the common adverse reactions of umbilical cord blood transfusion are increased body temperature, hemoglobinuria and DMSO side effects, and these adverse reactions can be adjusted by themselves and can be eliminated within 48 hours. Umbilical cord blood is rich in hematopoietic stem / progenitor cells, NK, regulatory T cells, and MSC can all have therapeutic effects on IRC to varying degrees, and the immune cells in cord blood are mostly naive, immature immune cells, Therefore, the incidence and severity of graft-versus-host disease (GVHD) after clinical application of unrelated umbilical cord blood are low, avoiding a series of complications and high costs caused by complex GVHD prevention and treatment technology. At the same time, regulatory T cells (Treg) in umbilical cord blood account for about 10% of all lymphocytes. They are a group of lymphocytes with negative regulatory immune responses. They usually play an important role in maintaining self-tolerance and avoiding excessive immune responses to damage the body. Function, its infusion can directly treat IRC. The number of NK cells in IRC patients is reduced, the immune monitoring effect is weakened, the homeostasis of the immune system cannot be maintained, and the immune cell function is hyperactive, leading to morbidity. However, CD16 + CD56 + NK cells are abundant in cord blood, and the amount of CD3 + T cells is the same as that in bone marrow. Most researchers believe that NK cells play an important role in immune surveillance in the body's immune system. They can regulate downstream immune cells by secreting cytokines or cytotoxicity, and thus play a protective role in autoimmune diseases. In addition, mesenchymal stem cells (MSC) contained in cord blood are another type of stem cells with high self-renewal and multi-directional differentiation potential, which can differentiate into a variety of tissue cells other than hematopoietic cells and have hematopoietic support , Immunomodulation, tissue repair and other functions are conducive to the restoration of bone marrow function in patients with hematopoietic disorders; at the same time, MSCs also have immunomodulatory, anti-inflammatory and tissue repair functions, which can reduce graft-versus-host disease (GVHD) and other transplant-related complications. Umbilical cord blood has the advantages of quick access, convenient source, no harm to donors, low HLA matching requirements, low incidence of graft-versus-host disease (GVHD) and low degree, making the clinical application of cord blood more and more widely , Its clinical treatment advantages have become increasingly prominent.

On May 1, 2009, the General Office of the Ministry of Health issued a notice on the first batch of the third category of medical technology that allows clinical application, clarifying that umbilical cord blood hematopoietic stem cell therapy technology is approved for clinical application as a third category of medical technology. In addition, the Technical Specification for Hematopoietic Stem Cell Transplantation clearly states that cord blood hematopoietic stem cells for clinical application should be provided by the cord blood hematopoietic stem cell bank approved by the National Health and Family Planning Commission. On July 4, 2019, the National Health and Welfare Commission issued a document that clearly stated that there are currently 7 cord blood hematopoietic stem cell banks that have passed the national acceptance practice, namely Shandong Bank, Beijing Bank, Tianjin Bank, Shanghai Bank, Zhejiang Bank, Guangdong Bank and Sichuan library.

This study intends to recruit IRIC patients, give cord blood infusion, observe its efficacy and safety, and detect changes in inflammation-related indicators before and after treatment. There are no relevant reports at China and abroad. This study can provide new treatment options for patients with IRIC. If it proves effective, it may rewrite the treatment guidelines for such diseases; in addition, this study may also provide a theoretical basis for expanding the application of cord blood in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years (adults, elderly), gender is not limited;

  * The diagnosis is definitely immune cytopenia (IRC), including autoimmune hemolytic anemia (AIHA, Hgb <100g / L, acquired pure red aplastic anemia (PRCA, Hgb <100g / L, EVANS syndrome ES, Hgb <100g / L and / or platelet count <30 × 109 / L, or cytopenia secondary to immune diseases (same treatment as before, or neutrophils <0.5 × 109 / L), at least after hormones If the treatment is not effective (PR has not been achieved after 4 weeks of hormone therapy) or cyclosporine 3-5mg / kg / d has not reached PR for half a year.

    * Those without abnormal cardiac function, abnormal liver function (total bilirubin 1.5 × ULN, ALT, AST≤3.0 × ULN), and abnormal renal function (serum creatinine≤1.0 × ULN) ④ ECOG score 0, 1 or 2; ⑤ Except autoimmunity There is no other secondary disease other than the disease; ⑥ Clearly understand the content of the trial, voluntarily participate in and complete this trial, and voluntarily sign an informed consent.

Exclusion Criteria:

* Age <18 years old or> 80 years old;

  * Patients with tumors (except carcinoma in situ); ③ Uncontrollable systemic infections or other serious diseases; ④ Women who are pregnant or lactating; ⑤ Patients with mental illness and potential impact Those with severe mental and mental illness who signed the informed consent form and followed up with the medical consultation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate Clinical remission rate Clinical remission rate Clinical remission rate: including CR and PR | 0.5~24 months
  Units of Measure %

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided